CLINICAL TRIAL: NCT01176084
Title: The Efficacy of a Low Carbohydrate Diet, With and Without Exercise, on Cardiovascular Disease Risk in Obese Men
Brief Title: Low Carb Diets & Exercise for Cardiovascular Disease (CVD) Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Dr Kathryn Hart, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lowcarbex_v1
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-07

CONDITIONS: Obesity
Keywords: low carbohydrate diet; obesity; moderate exercise; men
MeSH Terms: conditions — Obesity; Multiple Endocrine Neoplasia Type 1 | interventions — Diet, Carbohydrate-Restricted; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- low carbohydrate diet (Experimental)
  Interventions: Behavioral: low carbohydrate diet
- diet & exercise (Experimental)
  Interventions: Behavioral: low carbohydrate diet and exercise

INTERVENTIONS:
Behavioral: low carbohydrate diet
  Arms: low carbohydrate diet
Behavioral: low carbohydrate diet and exercise
  Arms: diet & exercise

SUMMARY:
The purposes of this study are:

To investigate the effects of a 6 month low carbohydrate diet in obese men on markers of heart health including blood fats, blood clotting factors, inflammatory markers and levels of body fat.

To investigate the added effect on heart health that regular moderate exercise may have when combined with a low carbohydrate diet in obese men.

ELIGIBILITY:
Inclusion Criteria:

* male
* 21-65 years
* body mass index (BMI) 27-40kg/m2
* not currently losing weight
* physically able to exercise at moderate intensity

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-01; Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
insulin levels

SECONDARY OUTCOMES:
body composition
lipid profile
body weight

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hiscutt, PhD, Principal Investigator — University of Surrey; Helen D Truby, PhD, Study Director — Monash University
Locations (1):
- Faculty of Health and Medical Sciences, University of Surrey, Guildford, Surrey, United Kingdom